# FEDERAL UNIVERSITY OF RIO GRANDE DO SUL SCHOOL OF MEDICINE GRADUATE PROGRAM IN HEALTH SCIENCES: GYNECOLOGY AND OBSTETRICS

# PERINEAL MASSAGE DURING LABOR FOR THE PREVENTION OF PERINEAL TRAUMA: A RANDOMIZED CLINICAL TRIAL

Project Number in CAAE: 77121923.5.0000.5327

PORTO ALEGRE 2024

# **Study Protocol**

# 1. Background and Rationale

Perineal trauma during childbirth, particularly episiotomy and spontaneous lacerations, is associated with pain, prolonged recovery, and complications during the puerperium. Evidence from prior meta-analyses (e.g., Aasheim et al., Cochrane 2017) suggests potential benefits of perineal massage in reducing these outcomes. This study aims to contribute robust evidence through a properly randomized, controlled design conducted in a high-volume public hospital.

# 2. Objectives

Primary Objective: To evaluate whether perineal massage reduces the incidence of intact perineum (absence of episiotomy or laceration) compared to standard care.

Secondary Objectives: To assess differences between groups in the degree of lacerations, need for sutures, incidence of episiotomy, neonatal APGAR scores, and second stage labor duration.

# 3. Study Design

Type: Interventional, Randomized Controlled Trial

Model: Parallel Assignment

Allocation: 1:1 (Massage vs. Control) Estimated enrollment: 466 participants

Location: Hospital de Clínicas de Porto Alegre (HCPA), Brazil

# 4. Eligibility Criteria

#### Inclusion:

- Women ≥18 years old

- Gestational age: 37-42 weeks

- Cephalic presentation
- First stage of labor
- No history of perineal massage in prenatal period

### **Exclusion:**

- Cesarean delivery
- Diagnosis of HELLP syndrome
- Unstable maternal or fetal vital signs

# Statistical Analysis Plan (SAP)

#### 1. Overview

The SAP describes the statistical methods that will be used to analyze the data from the trial and to address each primary and secondary objective.

# 2. Sample Size Calculation

Based on Cochrane meta-analysis by Aasheim et al. (2017), a reduction in episiotomy rate from 22% to 12% (RR = 0.55)

Power: 80%

Sample size: 466 participants (233 per arm)

# 3. Population for Analysis

Full Analysis Set (FAS): all randomized participants, analyzed by original assignment (intention-to-treat)

Per Protocol (PP): participants who adhered to the assigned intervention

#### 4. Statistical Methods

**Descriptive Statistics:** 

- Continuous variables: mean ± SD or median (IQR), depending on normality
- Categorical variables: frequency and percentage

# Test of Normality:

- Shapiro-Wilk test

# Between-Group Comparisons:

- Normal distribution: independent samples t-test
- Non-normal distribution: Mann-Whitney U test
- Categorical variables: Pearson Chi-square, Fisher's exact test, or Yates' correction

Within-Subject Comparisons (Pre/Post if applicable):

- Normal distribution: paired t-test
- Non-normal distribution: Wilcoxon signed-rank test
- Dichotomous categorical variables: McNemar test

#### Significance Threshold:

- Two-sided p-value ≤ 0.05 will be considered statistically significant.

# Missing Data:

- Assessed for patterns and handled using complete-case analysis or imputation if necessary.

#### 5. Software

Statistical analysis will be conducted using SPSS for Windows, version 18.0.